CLINICAL TRIAL: NCT01979679
Title: A D2 Receptor Occupancy and fMRI Study in Schizophrenic Subjects Treated With Lurasidone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Dainippon Sumitomo Pharma America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-6481
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lurasidone 80 mg per day (Active Comparator): Lurasidone 80 mg per day
  Interventions: Drug: Lurasidone 80 mg
- Lurasidone 120 mg per day (Active Comparator): Lurasidone 120 mg per day
  Interventions: Drug: Lurasidone 120 mg
- Lurasidone 160 mg per day (Active Comparator): Lurasidone 160 mg per day
  Interventions: Drug: Lurasidone 160 mg

INTERVENTIONS:
Drug: Lurasidone 80 mg
  Arms: Lurasidone 80 mg per day
Drug: Lurasidone 120 mg
  Arms: Lurasidone 120 mg per day
Drug: Lurasidone 160 mg
  Arms: Lurasidone 160 mg per day

SUMMARY:
The purpose of this research study is to measure how many of the dopamine receptors lurasidone occupies throughout the brain of patients with schizophrenia or schizoaffective disorder and over what time period the occupancy occurs. This is research because lurasidone is an investigational medication that has not yet been approved by the Food and Drug Administration (FDA). Dopamine receptors have key roles in many processes, including the control of motivation, learning, and fine motor movement. The degree of occupancy and the transience of occupancy D2 receptor occupancy for optimal clinical response and to prevent relapses is a controversial area that this study will address.

In this study Positron Emission Tomography (PET) scanning will be performed with D2/D3 ligand 18F-fallypride (a radioactive, injectable substance) to help the researchers measure the use of these receptors. Researchers hope that quantifying the amount of receptors being occupied by the medication will help them to determine the best dose of study medication in terms of improvement and least side effects related to body size and gender as well as in preventing relapse that may be related to hypersensitivity. Magnetic Resonance Imaging (fMRI) will also be performed. MRI is a scanning method which makes pictures of parts of the brain using a large magnetic field. This study will use a particular kind of MRI called fMRI, or functional MRI. fMRI takes pictures of the brain while the person is thinking or doing a simple task. fMRI will allow the researchers to investigate patients regional brain activation during cognitive (mental) and emotional tasks.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to participate in this study if they:

* are 18 to 60 years of age at the day of first dosing.
* are diagnosed with schizophrenia or schizoaffective disorder.
* are female, subject must be using an acceptable method of birth control or be surgically sterile or postmenopausal. Postmenopausal is defined as no period for at least 12 months. Acceptable methods of birth control include oral, injectable or implanted contraceptives, and barrier methods such as condoms, diaphrams, and spermicides.
* are able to provide written informed consent.
* can safety have an MRI (no metal in the body, not claustrophobic).

Exclusion Criteria:

Subjects are not eligible to participate in this study if they:

* are treatment resisitant or intolerant to lurasidone.
* have had extensive radiation exposure (the study doctor will discuss this with the subject).
* if they have tremors or shaking of the limbs.
* are pregnant or trying to become pregnant or breastfeeding.
* are colorblind.
* have a current or past history of a major medical illness or have abnormal lab values which the study doctor feels is significant (any abnormal lab values will be discussed with the subject).
* are taking certain medications. The study doctor will discuss these medicines with the subject.
* have a history of alcohol, cannabis or cocaine abuse within two weeks prior to the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-12; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
D2 receptor occupancy | Up to 6 weeks
  To determine whether additional D2 receptor occupancy can be accomplished with doses of 160 mg of lurasidone per day.

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Potkin, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Medical Center, Orange, California, United States

REFERENCES:
- [Result] Potkin SG, Keator DB, Kesler-West ML, Nguyen DD, van Erp TG, Mukherjee J, Shah N, Preda A. D2 receptor occupancy following lurasidone treatment in patients with schizophrenia or schizoaffective disorder. CNS Spectr. 2014 Apr;19(2):176-81. doi: 10.1017/S109285291300059X. Epub 2013 Sep 30. PMID 24073841